CLINICAL TRIAL: NCT01555359
Title: Telomerase Activity Of CD34+ Cells - Marker For Mobilization Quality And Predictor For Engraftment After Autologous Hematopoietic Cell Transplantation
Brief Title: Telomerase Activity as a Marker For Mobilization Quality
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: HCT-TEL-001
Record Dates: First submitted 2012-03-13; First posted 2012-03-15 (Estimated); Last update posted 2012-03-15 (Estimated); Status verified 2012-01

CONDITIONS: Lymphoma; Multiple Myeloma
MeSH Terms: conditions — Lymphoma; Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients undergoing stem cell collection

SUMMARY:
Autologous hematopoietic cell transplantation (HCT) is a treatment strategy used as advanced line therapy for different malignancies, mainly hematological. Its main advantage lies in the ability to provide hematologic and immune rescue after high dose chemotherapy therapy. The first requirement of a successful transplantation is recruitment of sufficient amount of cells. This is achieved by mobilizing CD34+ stem cells from the bone marrow to the peripheral blood, by G-CSF priming, and then harvesting the cells from the peripheral blood at the right timing by means of apheresis. Currently, the decision on the optimal collection timing is based on the pre-collection CD34 cells blood concentrations.

The investigators goal is to investigate whether telomerase, the telomere elongation enzyme, which constitutionally and solely expressed in progenitor cells, is correlated with collection and post HCT engraftment characteristics.

The investigators will collect blood from patients when starting GCSF and on the day of planned apheresis. Pearson correlation test will be used to correlate between telomerase activity in the samples and with collection and engraftment characteristics.

DETAILED DESCRIPTION:
Autologous hematopoietic cell transplantation (HCT) has revolutionized the curative approach to a number of malignancies by providing hematopoietic and immune rescue after high dose cytoreductive therapy. In cases of residual disease, patients are usually treated with chemotherapy to repress the disease, thereafter G-CSF injections are given serially to encourage stem cell proliferation in the bone marrow and mobilization of the stem/progenitor cells to the peripheral blood. Another approach, usually utilizes in myeloma patients is the administration of G-CSF in steady state (without administration of chemotherapy) and consequently collection of the CD34+ cells.

The minimum number of CD34+ cells threshold requires for HCT is currently defined as 2 x 10^6/kg. However, the optimal dose in terms of engraftment may be even higher (>5x10^6/kg), especially when platelet recovery is considered.

In clinical practice, the right timing for collection is decided upon measurement of CD34, a membrane glycoprotein of progenitors and stem-cells. CD34 levels are measured in the expected maximal effect of the G-CSF priming, and accordingly the collection is scheduled. Practically, if the circulating CD34+cell count is ≥20/μL, 90% of collections performed the following day would be expected to yield ≥2.0x106 CD34+cells/kg (Gordon, BMT 1997). However, in cases higher doses of CD34+ cells are required (e.g. for tandem HCT), CD34+ threshold may not be sufficient to determined collection yield.

G-CSF based mobilization regimens have a 5-30% failure rate amongst patients, however in patients with risk factors, up to 60% of the patients are failed to mobilize. Poor mobilization has significant consequences for the patient with potential loss of transplantation as a treatment option. Repeated attempts at mobilization increase resource utilization, morbidity and patient inconvenience. Therefore attempts to identify patients who would mobilize poorly are of clinical significance.

Human telomerase, a unique ribonucleoprotein complex, is inactive in normal somatic cells but present in high levels in more than 90% of all malignancies. The enzyme, synthesize new telomeric repeats at the 3' ends of chromosomes.

As oppose to other normal cells, stem cells are unique in that they carry active telomerase which provides them with longer life span. Previous study from our lab showed that in patients and healthy donors, the administration of GCSF was associated with a 14th fold increase of telomerase activity levels in peripheral blood CD34+ cells.

Working hypothesis:

Telomerase activity in mobilized stem cells is correlated with both the absolute number of the collected cells and with the quality of the future engraftment after high dose therapy and HCT

Specific aims:

1. To investigate the correlation between telomerase activity of CD34+ cells in the day of collection and the total number of collected CD34+ cells in a cohort of 50 patients undergoing stem cells mobilization and collection.
2. To explore the association between telomerase activity of CD34+ cells and the engraftment characteristics (time to platelets>50000/microL, time to platelets>150000/microL, time to neutrophils>500/microL, time to neutrophil>2000/microL).
3. To develop an algorithm based on CD34+ cells levels and CD34+ telomerase activity, both measured on the day of collection, that can serve as predictor for the total number of CD34+ cells to be collected.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years
2. Patient is candidate for stem cell mobilization and collection
3. Patient is willing to sign an informed concent

Exclusion Criteria:

1. Age <18 years
2. Patient not willing or not in a state to sign an informed concent
3. Pregnant women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing stem cell mobilization and collection
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2012-02; Study Completion 2013-02 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Ron Ram, M.D., Principal Investigator — BMT Unit, Davidoff Cancer Center, Rabin Medical Center, Beilinson Hospital
Locations (1):
- BMT Unit, Davidoff Cancer Center, Rabin Medical Center, Beilinson Hospital, Petah Tikva, Israel

REFERENCES:
- [Background] Szyper-Kravitz M, Uziel O, Shapiro H, Radnay J, Katz T, Rowe JM, Lishner M, Lahav M. Granulocyte colony-stimulating factor administration upregulates telomerase activity in CD34+ haematopoietic cells and may prevent telomere attrition after chemotherapy. Br J Haematol. 2003 Jan;120(2):329-36. doi: 10.1046/j.1365-2141.2003.04043.x. PMID 12542495